CLINICAL TRIAL: NCT04287959
Title: Randomised Control Trial Comparing High Flow Weaning Strategies for Infants With Bronchiolitis: Pilot Study
Brief Title: SWISH Trial (Strategies for Weaning Infants on Supportive High Flow)
Acronym: SWISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/OCT/7769
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Disease; Bronchiolitis, Viral; Infant Morbidity
MeSH Terms: conditions — Respiration Disorders; Bronchiolitis, Viral

STUDY DESIGN:
Intervention Model Description: Given this is a pilot study, a recruitment target has not been set. Instead the study will aim to assess recruitment success which will inform a larger multicentre trial if deemed feasible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: wean to 30% (Active Comparator): wean to 30% oxygen on high flow and then turn off high flow support and place onto standard low flow oxygen.
  Interventions: Device: High flow nasal cannula support
- B: wean to 21% (Active Comparator): wean to 21% oxygen on high flow and then turn off high flow support and place directly into air.
  Interventions: Device: High flow nasal cannula support

INTERVENTIONS:
Device: High flow nasal cannula support — airvo2 highflow devices will be used.

SUMMARY:
Bronchiolitis is a common type of chest infection that tends to affect babies and young children under a year old. In older children and adults, the same viruses that cause bronchiolitis lead to the 'common cold'.

The symptoms of bronchiolitis are like a common cold and include a blocked or runny nose, a cough and a mildly raised temperature.

Bronchiolitis affects the bronchioles which are the smaller breathing tubes in the lungs. They produce more mucus than usual and become swollen, leading to a cough and a runny nose. In more severe cases, the tubes become clogged up with mucus which causes breathing problems.

In some babies, the breathing problems may present as breathing fast, with in-drawing of the muscles around the rib cage, and in rare cases, very young babies with bronchiolitis may stop breathing for brief periods ('apnoea'). The illness usually starts with a mild runny nose or cough, gets worse over three to five days or so, and then slowly gets better, usually lasting about 10 to 14 days in total.

Around 2 in 100 infants with bronchiolitis will need to spend some time in hospital during the course of their illness. This is usually for one of two reasons: they need oxygen treatment to keep their oxygen saturations within acceptable levels or they cannot manage to feed from the breast or a bottle because of a blocked nose or difficulty breathing.

Here at the Children's Hospital for Wales we are using 'High flow' to deliver oxygen. This is a relatively new concept on the general paediatric wards, and more established in a setting such as High Dependency Unit (HDU). However, we have been using it successfully on the wards for the last 3 years.

High flow device delivering a mixture of oxygen and air at high flow to help open the child's airways so that their lungs can add oxygen to their blood. It is given through a set of prongs (short plastic tubes) inserted just inside the nostrils.

Research has shown that the early use of high flow can reduce the chances of the child needing escalation of care to a high dependency unit or paediatric intensive care unit.

The investigators are interested in studying the process of weaning high flow support once the child is over the worst of their illness. This will enable the investigators to use the most effective method of weaning babies from their high flow, and ready for discharge. This has the potential to reduce the number of hours spent in hospital for babies and their parents or guardians.

DETAILED DESCRIPTION:
Bronchiolitis is the commonest respiratory infection in infancy leading to hospital admission. 46 per 1000 infants were admitted to hospital with bronchiolitis in England in 2011 and more recent studies suggest this number has remained static. This has a significant cost burden on the NHS. Respiratory support, mainly oxygenation, and keeping infants well hydrated are the mainstay of management in hospital.

Respiratory support has traditionally been the domain of intensive care settings. This has been provided through an escalation of therapy from simple oxygen delivery by nasal cannula, to non-invasive ventilation with Continuous Positive Airway Pressure (CPAP) and finally to intubation with mechanical ventilation. These latter two strategies require highly skilled staff, so are costly, and are associated with a greater incidence of adverse events including ventilator-induced lung injury, barotrauma, and potential neurotoxicity associated with sedation. Over the last decade High Flow Nasal Cannula (HFNC) therapy has emerged as a new method to provide respiratory support for bronchiolitis. HFNC therapy works by delivering an increased volume of air and oxygen into the nasal passages than standard sub-nasal oxygen therapy, using a higher flow of humidified and heated gas. These increased flow rates exceed peak inspiratory flow and thereby result in more efficient delivery of oxygen to the terminal airways. Physiological studies have demonstrated reduced work of breathing and improved gas exchange. The PARIS study has demonstrated that HFNC can be used in a ward setting to reduce admission rates to the Paediatric Intensive Care Unit (PICU). 12% of the study population receiving HFNC needed escalation to PICU compared to 23% receiving standard care (oxygen therapy). The safety data from the PARIS study shows no difference in adverse effects between HFNC and standard oxygen therapy. Numerous studies over the last three decades have investigated the role of various medications in managing infants with bronchiolitis including adrenaline, steroids, salbutamol, and hypertonic saline; none of these studies have definitively changed the outcome of the disease nor the length of stay in hospital. Although the PARIS study showed a reduction in number of patients requiring escalation of care, it did not demonstrate any difference to the total length of stay in hospital.

Aim Since HFNC is a relatively new method of providing respiratory support in bronchiolitis, there is lack of evidence on weaning strategy. The investigators primary aim is to examine the feasibility of different weaning strategies for infants, up to 12 months of age, supported on HFNC for bronchiolitis. The secondary outcomes include the time from decision to wean HFNC to the patient no longer requiring respiratory support and a safety assessment of the weaning strategies. This may lead to shorter total length of stay in hospital, without compromising their care. Infants with bronchiolitis who are on HFNC (the devices used will be Airvo 2, Fisher & Paykel Healthcare) will be on a flow of 2L/kg/min (maximum 20L/min) and variable oxygen concentration to maintain target oxygen saturations >90%. The participants will be randomised into one of two arms for weaning a) titrating oxygen to FiO2 21% and then stopping HFNC b) titrating oxygen to FiO2 30% and switching HFNC to low flow oxygen.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of bronchiolitis
* Age >4 weeks and <12 months
* Needs HFNC respiratory support in a ward setting for more than 12 hours

Exclusion criteria:

* Requirement for imminent intubation and ventilation or having received mechanical ventilation during the current hospital admission
* Requirement for imminent CPAP support
* Pre-existing or concomitant, non-viral respiratory infection
* Pre-existing respiratory disease
* Ready to wean high-flow after <12 hours of its initiation
* Weight >10kg
* Low level of consciousness
* Apnoeas*
* Cyanotic heart disease
* Basilar skull fracture
* Upper airway obstruction
* Craniofacial malformations
* Infants on home oxygen
* Ex-premature infants (born at <32 weeks gestation)

Ages: 4 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Examine the feasibility of different weaning strategies for infants with bronchiolitis requiring HFNC. | This will be during the recruitment time of the study (2 years)
  we will assess the following objective in this feasibility trial:
  • identify the proportion of eligible patients approached who consent to the study; We will use a traffic light system to determine progress to a multi-centre RCT.
Identify the proportion of recruited patients who supply secondary outcome data. | This will be during the recruitment time of the study (2 years)
  We will assess the following objective:
  identify the proportion (percentage) of recruited patients who supply primary outcome data(time spent in hospital).
Assess the adherence of the teams on the ward to the weaning protocol assigned during randomisation. | This will be during the recruitment time of the study (2 years)
  We will assess the following objective:
  to review the adherence to the weaning protocol assigned during randomisation, in particular if this can be complied with in a ward setting with a large number of healthcare staff. This will be measured as a yes or no response and calculated as a percentage/proportion.
Assess the acceptability of HFNC and the weaning strategy by parents and healthcare staff. | This will be during the recruitment time of the study (2 years)
  We will assess the following objectives:
  to assess the acceptability of HFNC and the weaning strategy by parents and healthcare staff via questionnaires only.

SECONDARY OUTCOMES:
Time taken to wean off the highflow machine as measured in minutes and hours. | This will be during the recruitment time of the study (2 years)
  The main secondary outcome is the comparison of time taken from the patient being ready to wean HFNC to discontinuing any respiratory support. This will be measured in minutes and hours and a comparison made between the two intervention arms.
To assess the safety of the different weaning strategies used. | This will be over the 2 years of recruitment time of the study.
  The safety outcome measures comprise the following:
  * rates of failure to wean strategy (defined as fulfilment of the 'failure to wean criteria' which results in a patient becoming temporarily ineligible for oxygen weaning);
  * rates of respiratory escalation requiring CPAP or invasive ventilation (proportions);
  * rates of air leaks and other morbidities such as pnuemothorax or muscosal injury (proportions);
  * readmission rates within 14 days of discharge from hospital
  * mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Edwards, PhD, BM, Principal Investigator — CAVUHB
Locations (1):
- Children's Hospital for Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Towriss C, Dafydd C, Edwards M. High-flow weaning strategies for infants with bronchiolitis: protocol for a pilot randomised controlled trial in the UK. BMJ Open. 2024 Nov 9;14(11):e087672. doi: 10.1136/bmjopen-2024-087672. PMID 39521467